CLINICAL TRIAL: NCT02093000
Title: A Multicenter, Prospective, Non-interventional Study of Maintenance Avastin® (Bevacizumab) Following Induction Treatment With Platinum Doublet Plus Avastin® in Patients With Advanced Lung Adenocarcinoma
Brief Title: A Study Examining Maintenance Bevacizumab (Avastin®) Monotherapy in Participants With Advanced Lung Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29261
Record Dates: First submitted 2014-03-19; First posted 2014-03-20 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Lung Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — Bevacizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Bevacizumab: Participants who have received the induction phase of 4-6 cycles of bevacizumab plus platinum doublet chemotherapy will be treated with bevacizumab as maintenance treatment, according to approved label and local reimbursement.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Participants will receive bevacizumab 7.5 milligrams per kilograms (mg/kg) intravenously according to bevacizumab summary of product characteristics/local labeling.
  Other Names: Avastin®

SUMMARY:
This prospective, open-label, single arm, non-interventional study will investigate the effectiveness of bevacizumab monotherapy in participants with lung adenocarcinoma who previously received 4 to 6 cycles of induction platinum doublet plus bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Participant who previously received 4 to 6 cycles of induction platinum doublet plus bevacizumab
* Participant who received only 1 cycle of bevacizumab maintenance treatment
* Meet summary of product characteristics guidelines

Exclusion Criteria:

* Participant who received the first cycle of maintenance bevacizumab more than 4 weeks after the postinduction tumor assessment
* Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving Avastin monotherapy as maintenance treatment
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2014-11-30 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS), Defined as Time From First Dose of Maintenance Avastin Treatment Until Disease progression or death from any cause | Baseline up to 40 months

SECONDARY OUTCOMES:
PFS, defined as time from first dose of induction Avastin treatment until disease progression or death from any cause | Baseline up to 40 months
1-year overall survival defined as time from first dose of induction Avastin treatment until death from any cause | 12 months
Percentage of participants by best overall response | Baseline up to 40 months
Percentage of participants with adverse events | Baseline up to 40 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (16):
- Hungary (16):
  - Orszagos Koranyi TBC es Pulmonologiai Intezet, Budapest
  - Semmelweis Egyetem X; Pulmonologiai Klinika, Budapest
  - Uzsoki Utcai Korhaz, Budapest
  - Debreceni Egyetem, Klinikai Kozpont, Tudogyogyaszati Klinika, Debrecen
  - Csongrad Megyei Mellkasi Betegsegek Szakkorhaza, Deszk
  - Veszprem Megyei Onkormanyzat Tudogyogyintezet, Farkasgyepű
  - Petz Aladar Megyei Oktato Korhaz, Győr
  - Bekes Megyei Tudokorhaz; I. Tudobelosztaly, Gyula
  - Bacs-Kiskun Megyei Korhaz, Kecskemét
  - Matrai Gyogyintezet, Mátraháza
  - Szabolcs-Szatmar-Bereg County Josa Andras Hospital; 1St Depatment of Pulmonary Medicine, Nyíregyháza
  - University of Pecs; 1St Department of Medicine, Pécs
  - Fejer Megyei Szent Gyorgy Korhaz, Székesfehérvár
  - Vas Megyei Markusovszky Korhaz ; Oncoradiology, Szombathely
  - Komárom-Esztergom Megyei; Szent Borbála Kórháza, Tatabánya
  - Tudogyogyintezet Torokbalint, Törökbálint